CLINICAL TRIAL: NCT06768463
Title: Cytoreductive Gastrectomy After Systemic Therapy Versus Systemic Therapy Alone For Limited Metastasis Gastric Cancer: An Open-label Randomized Controll Trial
Brief Title: Cytoreductive Gastrectomy After Systemic Therapy Versus Systemic Therapy Alone For Limited Metastasis Gastric Cancer
Acronym: CYGAS-GC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYGAS-GC
Record Dates: First submitted 2024-12-26; First posted 2025-01-10 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Gastric Cancer; Gastric Cancer; Systemic Therapy; Cytoreductive Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Cytoreductive Gastrectomy After Systemic Therapy For Limited Metastasis Gastric Cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cytoreductive Gastrectomy After Systemic Therapy (Experimental): After 4 cycles of systemic therapy, the patients with complete response, or partial response, or stable disease undergo gastretomy.
  After gastrectomy, the patients continue to use systemic therapy.
  Interventions: Procedure: Cytoreductive Gastrectomy
- Systemic Therapy Alone (No Intervention): The patients only use systemic therapy.

INTERVENTIONS:
Procedure: Cytoreductive Gastrectomy — The patients undergo gastrectomy after 4 cycles of systemic therapy
  Arms: Cytoreductive Gastrectomy After Systemic Therapy

SUMMARY:
The results of the current studies to determine the optimal strategy for metastatic gastric cancer remain contrversial worldwide.

Hypothesis: Cytoreductive Gastrectomy After Systemic Therapy will improve survival time for metastasis gastric cancer compared to Systemic Therapy alone.

DETAILED DESCRIPTION:
Stomach cancer in Vietnam is often detected at a late stage, with about 30% of patients having distant metastases within the abdomen at the time of diagnosis. The optimal treatment choice for patients at this stage remains unclear. For cases with distant metastases within the abdomen, such as liver metastasis, peritoneal metastasis, or lymph node metastasis along the aorta (16a2/b1), systemic therapy remains the standard treatment unless there are complications such as bleeding or pyloric stenosis. Survival time for these cases is generally less than 1 year according to previous studies. However, with advances in gastric cancer treatment, many recent studies show a significant improvement in the survival of this group. According to the results of the Regatta study, the median survival time was 16.6 months for patients receiving only chemotherapy and 14.3 months for those undergoing gastrectomy followed by chemotherapy. This is the largest randomized comparative study to date comparing the efficacy of chemotherapy alone versus gastrectomy followed by chemotherapy. The study results showed that gastrectomy did not significantly improve survival for patients. Therefore, according to current treatment guidelines of the Japanese Gastric Cancer Association or the European guidelines, systemic systemic therapy remains the recommended option for cases of gastric cancer with intra-abdominal metastases.

However, according to the authors of the Regatta study, after a longer follow-up period and a more detailed analysis of the relationship between overall survival and the characteristics of gastric cancer, it was found that for lower third gastric cancer, gastrectomy had better survival outcomes compared to chemotherapy alone. For middle third gastric cancer, survival outcomes were equivalent between the two groups, while for upper third gastric cancer, total gastrectomy had worse survival outcomes compared to chemotherapy alone. This difference is explained by the fact that after total gastrectomy, the patient's general condition deteriorates, making it impossible to tolerate postoperative chemotherapy. Therefore, for advanced-stage gastric cancer, many studies recommend preoperative systemic therapy to increase drug tolerance, increase the rate of R0 resection, and improve survival. The JCOG 0605 study for bulky lymph node or para-aortic lymph node metastatic gastric cancer showed that preoperative chemotherapy helped achieve an R0 resection rate of 82%, with 3-year and 5-year survival rates of 59% and 53%, respectively, which were better than expected. Additionally, many other studies on the treatment of metastatic gastric cancer have also shown the effectiveness of neoadjuvant systemic therapy combined with gastrectomy and postoperative systemic therapy. The CONVO-GC-1 multicenter retrospective study in Japan, South Korea, and China with 1206 cases of metastatic gastric cancer who underwent gastrectomy after neoadjuvant systemic therapy showed an overall median survival of 36.7 months, with median survival for R0, R1, and R2 resection groups being 56.6 months, 25.8 months, and 21.7 months, respectively. This result shows that preoperative systemic therapy combined with gastrectomy and postoperative systemic therapy has the potential to improve survival for advanced-stage gastric cancer patients.

Additionally, studies on targeted therapy have also shown effectiveness in the treatment of advanced gastric cancer, improving patient survival. The randomized multicenter ToGA study conducted in 24 major hospitals worldwide showed that Trastuzumab combined with systemic therapy was effective in improving survival for metastatic gastric cancer compared to systemic therapy alone, with median survival times of 13.8 months versus 11.1 months (HR = 0.74; 95% CI: 0.60-0.91; p = 0.0046). Other studies on this topic have shown similar results, so currently, Trastuzumab combined with systemic therapy is recommended as the first choice for metastatic gastric cancer expressing Her 2.

The results of the above studies form the basis for current research trends at many major centers worldwide to determine the optimal strategy for metastatic gastric cancer, which remains an open question. Whether to choose systemic therapy as per current treatment guidelines or to combine systemic therapy with gastrectomy is still a question that requires more robust evidence for a definitive answer. Therefore, we conducted this study to determine the effectiveness of preoperative systemic therapy combined with gastrectomy and postoperative systemic therapy compared to systemic therapy alone for metastatic gastric cancer with the following research questions:

1. Does the combination of neoadjuvant systemic therapy, gastrectomy, and adjuvant systemic therapy improve survival time for metastatic gastric cancer compared to systemic therapy alone?
2. Is gastrectomy after neoadjuvant systemic therapy safe?

ELIGIBILITY:
Inclusion criteria General criteria

* Age 18-75
* GCLM detected on surgical exploration and demonstrated by histology or cytology
* Localized peritoneal carcinomatosis (P1 or P2 score), according to the classification of the Japanese Research Society for Gastric Cancer
* Liver metastasis lesions of maximum diameter ≤5 cm
* Para-aortic lymph node metastasis below the coeliac axis or above the inferior mesenteric artery (lymph node 16a1/b2 of maximum diameter≥1cm)
* Bilateral or unilateral Krukenberg tumors were allowed and considered 1 incurable organ site
* The accepted patient has two metastases
* Baseline Eastern Cooperative Oncology Group (ECOG) performance status < 1
* Basic laboratory tests demonstrating adequate bone marrow function (neutrophil count > 1500mm3, haemoglobin > 8g/dL, platelet count > 100,000/mm3), adequate liver function (bilirubin, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within upper limits of normal), adequate renal function (serum creatinine within the upper limit of normal)
* Expected survival > 3 months
* Able to tolerate enteral nutrition and adequate mental capacity to give informed consent
* Completed 4 cycles of first-line standard-of systemic therapy
* Repeat diagnostic laparoscopy after first-line treatment prior to randomization demonstrating feasible resection.

Eligibility criteria for resection & extent of proposed resection

* Staging scans (cross-sectional imaging) demonstrating no extra metastases (lung, bone,...)
* Cross-sectional imaging demonstrating no local progression of PM
* PCI score <12
* Cytology +ve alone (no gross PM) permissible for enrolment
* Feasible R0 resection (reasonable chance of negative margins on histology)
* Feasible D1, D1+ or D2 lymphadenectomy

Exclusion criteria

* Any extra-abdominal metastasis at diagnosis or during systemic treatment.
* Past history of malignancy other than gastric cancer diagnosed in the last 5 years except for basal cell carcinoma of skin or preinvasive cancer of cervix
* Patients in the reproductive age who declined to use an adequate means of contraception
* Significant disease or conditions which, in the investigator's opinion, would exclude patient from the study
* Uncontrolled concurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
* Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and lactating females
* Prior surgical treatment for GC involving resection
* Clinical or radiological progression during 1st line systemic treatment

  * Patients with radiological progression of LM (determined by RECIST criteria) to be excluded as disease is likely not responding well to 1st line treatment.
  * Patients with clinical progression of LM as defined by increasing ascites requiring intervention (ascitic tap/drain, hospital admission etc) or causing significant symptoms to the patient (tense distended abdomen, early satiety, shortness of breath etc).

    * Ascites volume as a reflection of disease control is difficult to assess and quantify or a reflection of disease progression. (15)
* Any patient deemed unresectable or requiring extensive resection beyond procedure approved in the study protocol

  * PCI > 12
  * Extensive bowel / mesentery involvement requiring >2 separate / non-contiguous small or large bowel resections in addition to the gastrectomy
  * Involvement of the head of pancreas or bile duct
  * PM or nodal disease in the hepatoduodenal ligament
  * Involvement of major vascular structures
  * Involvement of esophagus precluding a reasonable chance of R0 resection by transhiatal approach Withdrawal Criteria
* Patient decides to withdraw from the study, or
* The investigator concludes that it is in the patient's best interest to discontinue study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-07-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Median survival time | 36 months after surgery
  the median length of time from the date of randomization to death from any cause or to the last follow-up for a surviving patient the median length of time from the date of randomization to death from any cause or to the last follow-up for a surviving patient
Progression-free survival (PFS) | 3 year after surgery
  Time interval from randomization to either radiological/clinical recurrence (Arm 1) or progression (Arm 2) or death from any cause. Patients who remained alive and without recurrence at the time of analysis or who are lost to follow-up will be censored at the date last seen

SECONDARY OUTCOMES:
Overall survival (OS | 3 year after surgery
  the time interval from randomization to death from any cause. Patients who remained alive at the time of analysis or who are lost to follow-up will be censored at the date last seen and intention-to-treat analysis will be performed
Cytoreductive completenes of peritonectomy (for Arm 1) | within 30 days after surgery
  The compleness of peritonectomy
  * CC-0: no peritoneal seeding visualized within the operative field
  * CC-1 indicates nodules persisting after cytoreduction less than 2.5 cm
  * CC-2 has nodules between 2.5 and 5 cm
  * CC-3 indicates nodules greater than 5 cm or a confluence of unresectable tumor nodule at any site within the abdomen or pelvis.
R0 resection rate (for Arm 1) | 3-month after conversion surgery
  Percentage of cases achiving R0 resection after cytoreductive surgery.
  Curability after conversion surgery (R0/R1/R2) defined as:
  * R2 surgery: macroscopically positive residual tumor at margins, invasive lesion, other metastatic lesions; or cytoreductive completeness of 1-3 when performing peritonectomy
  * R1 surgery: no R2 criteria; microscopically positive margins, or positive cytology lavage after gastrectomy, or finding of malignant lesion in the 3-month postoperative imaging
  * R0 surgery: no R1 or R2 surgery, and no finding of malignant lesion in thẻ 3-month postoperative imaging
Early complication rate (Arm 1) | 30-day postoperative
  Rate of any complications happened intraoperative and 30-days post-operative, classified by Clavien - Dindo classification
Late comlication rate (Arm 1) | 3 year after surgery
  Rate of any complications happened after 30-days postoperative, classified by Clavien - Dindo classification
Pathological response rate (Arm 1) | 30-day postoperative
  proportion of patients achieving grade 2 or more according to the histological criteria of the Japanese Classification of Gastric Carcinoma
Length of post-operative hospital stay | 30-day postoperative
  Time from day of surgery until day of discharge
Quality of life Quality of life Quality of life | 1 year after surgery or after chemotherapy
  The European Organization for Research and Treatment (EORTC) of Cancer quality of life questionnaire (EORTC-QLQ C30)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No